CLINICAL TRIAL: NCT02980146
Title: Correlation Between HLA-E Overexpression by Tumor Cells and the Biology of Tumor-infiltrating Lymphocytes Depending on the Microsatellite Status in Colorectal Cancer.
Brief Title: Impact of HLA-E Overexpression by Tumor Cells on the Biology of TIL in Colorectal Cancer
Acronym: HLA-E CCR
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: U892 INSERM Team 3 (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC16_0212
Record Dates: First submitted 2016-11-21; First posted 2016-12-02 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: ColoRectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 mL of Blood, a tumor fragment and a fragment of colonic mucosa
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group "patients with colorectal cancer": Major patients treated surgically for colorectal cancer at Nantes University Hospital or at the Institut de Cancerologie de l'Ouest and agreeing to participate in the study
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study

SUMMARY:
Accumulating evidences suggest that colorectal cancer (CRC) progression is not solely determined by the genetic abnormalities of the tumor cells but also by the host response. Indeed, recent studies in CRC have associated improved survival with a high number of tumor-infiltrating (TIL) memory and cytotoxic T lymphocytes, suggesting a link between tumor progression and in situ T cell response. Gene expression profiling studies have clearly isolated a well-known subgroup of CRC characterized by microsatellite instability (MSI) CRC, associated with a strong immune response signature involving both Th1/cytotoxic and immune evasion pathways. Moreover, the investigators have previously shown that HLA-E/β2m is overexpressed by tumor cells in roughly 20% of CRC and is associated with a worse prognosis, most likely due to NK and T effector cell functions upon engagement with the inhibitory NK receptor CD94/NKG2A. However, our recent results on an enlarger cohort of patients suggest that if this observation holds true for MSS CRC, HLA-E over-expression is inversely associated with a good prognosis in MSI CRC. Thus, the phenotype and function of TIL, depending on the MSI/MSS status of CRC have to be precised. The investigators hypothesized that in MSI CRC, known to express a high number of MSI-H related frameshift peptides which represent a pool of tumor specific antigens, HLA-E could present peptides to TCR of non conventional CD8+ HLA-E-restricted alpha-betaT cells (also expressing CD94), then inducing a strong antitumor cytolytic activity. Therefore, the aim of this project is to determine the exact phenotype, function and specificity of the CD94+ TIL in CRC, depending on both the HLA-E and the MSI/MSS status of tumor cells. These results could impact the clinical practice as anti-NKG2A monoclonal antibodies or frameshift peptide based immunotherapy that could be promising new therapeutic options in CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Major patients treated surgically for colorectal cancer at the Nantes University Hospital or the West Institute of Cancerology
* Patients agreeing to participate in the study

Non inclusion Criteria:

* Age> 85 years
* Neoadjuvant or immunosuppressive therapy for other pathology
* Size of the tumor insufficient to carry out all the samples dedicated to the research without constraining the diagnostic step (tumoral sampling at least equal to 1 cm3)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients treated surgically for colorectal cancer at the Nantes University Hospital or the West Institute of Cancerology
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-06-01; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
The phenotype of TIL will be precised by immunohistochemisry and flow cytometry using various combinations of monoclonal antibodies to identify different subset of TIL and their frequency, especially those expressing NKG2A or NKG2C chain. | Until 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Céline BOSSARD, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No